CLINICAL TRIAL: NCT03319524
Title: Prospective Open Label Clinical and Genetic Testing of Patients With Usher Syndrome
Brief Title: Clinical and Genetic Testing of Patients With Usher Syndrome
Status: Completed | Type: Observational
Sponsor: Sensor Technology for Deafblind (Industry)
Collaborators: Burnasyan Federal Medical Biophysical Center (Other Government); Scientific and Clinical Center for Otorhinolaryngology of FMBA of Russia (Unknown); Federal State Budgetary Institution Research Center for Medical Genetics (Unknown); ANO Laboratory Sensor-Tech (Unknown); Oftalmic LLC (Unknown); Deaf-Blind Support Foundation Con-nection (Unknown)
Responsible Party: Sponsor
Other Study IDs: RU-USH-09-2016
Record Dates: First submitted 2017-10-02; First posted 2017-10-24 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Usher Syndrome; Congenital Deafness; Retinitis Pigmentosa
MeSH Terms: conditions — Usher Syndromes; Retinitis Pigmentosa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is aimed to characterize Russian population of Usher patients.

DETAILED DESCRIPTION:
This study is aimed to characterize Russian population of Usher patients.

Tasks:

Stage 1. Formation of the primary cohort of patients. Patients pre-recruiting will be performed based on Deaf-Blind Support Foundation "Con-nection" patient database analysis. Patients with clinically confirmed Usher syndrome will be evaluated according to available data of the clinical examination.

Stage 2. Clinical examination of patients.

Each patient will undergo the following diagnostic procedures according to the unified protocol:

* Visometry (with correction and without correction)
* Ophthalmoscopy
* Perimetry
* Optical coherence tomography
* Electroretinography
* Visually evoked potentials
* Refractometry
* Pneumotonometry
* Biomicroscopy
* Tonal audiometry
* Electronic audiometry (ASSR test)
* Acoustic impedance measurement
* Vestibulometry
* Electronystagmography
* Any additional examinations and consultations if necessary

Medical record will be developed and maintained for each patient consisting results of extended clinical examination.

Stage 3. Genetic study of patients. All enrolled patients will undergo single 4 ml peripheral venous blood sampling. DNA will be extracted from leucocytes. DNA samples will be analyzed and placed for long-term storage in liquid nitrogen. Statistical and bioinformatic analysis of detected genetic mutations in the study cohort will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patient fulfill the clinical characteristics for Usher syndrome type I, II or III as defined by the Usher syndrome consortium
* According to the results of audiometry, hearing loss is moderate or severe (level of acoustic threshold of audibility is 41 decibel and higher).
* Results of perimetry for each eye show narrowing for 15 degrees or more.
* Patient is familiar with Participant information sheet
* Patient signed informed consent form

Non-inclusion Criteria:

* Participation in other clinical trials (or administration of investigational drugs) during 3 months prior inclusion
* Any conditions limiting compliance (dementia, neuropsychiatric disease, drug and alcohol abuse etc.)
* Medical history of traumatic injury of eyes, barotrauma, concussion, craniocerebral trauma, cerebrovascular accident

Exclusion Criteria:

* Patient's refusal from the further participation in the trial
* Decompensated diabetes mellitus
* Severe coronary artery disease
* Chronic infectious disease
* Patients with malignant tumors including postoperative period, patients receiving chemotherapy and/or radiotherapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is assumed that at least 28 patients of the Russian population of men and women aged 18 to 65 years, with verified diagnosis of Usher syndrome (type I, II or III as defined by the Usher syndrome consortium), will take part in this research study.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Changes in visual acuity | Up to 4 weeks
  Measured by visometry
Changes in structures of fundus of the eye-1 | Up to 4 weeks
  Measured by ophthalmoscopy
Changes in structures of fundus of the eye-2 | Up to 4 weeks
  Measured by optical coherence tomography
Changes in visual field | Up to 4 weeks
  Measured by perimetry
Changes in retinal ganglion cell dysfunction | Up to 4 weeks
  Measured by electroretinography
Changes in brain visual cortex neural pathways | Up to 4 weeks
  Measured by visually evoked potentials
Changes in optical refraction | Up to 4 weeks
  Measured by refractometry
Changes in intraocular pressure | Up to 4 weeks
  Measured by pneumotonometry
Changes in the lens, cornea, anterior segment of the eye | Up to 4 weeks
  Measured by biomicroscopy
Changes in hearing-1 | Up to 4 weeks
  Measured by tonal audiometry
Changes in hearing-2 | Up to 4 weeks
  Measured by electronic audiometry (ASSR test)
Changes in efficient sound transmission in the middle ear | Up to 4 weeks
  Measured by acoustic impedance measurement
Changes in vestibular functions | Up to 4 weeks
  Measured by vestibulometry
Changes in vestibular reactions | Up to 4 weeks
  Measured by electronystagmography

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir N Trubilin, MD, PhD, Prof, Principal Investigator — State Research Center Burnasyan Federal Medical Biophysical Center Federal Medical-Biological Agency
Locations (6):
- Russia (6):
  - Federal State Budgetary Institution "Research Center for Medical Genetics", Moscow
  - Deaf-Blind Support Foundation "Con-nection", Moscow
  - State Research Center Burnasyan Federal Medical Biophysical Center Federal Medical-Biological Agency, Moscow
  - Scientific and Clinical Center for Otorhinolaryngology of FMBA of Russia, Moscow
  - Oftalmic LLC, Moscow
  - Autonomous nonprofit organization "Scientific and industrial laboratory "Sensor technology for deafblind", Moscow

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ivanova ME, Trubilin VN, Atarshchikov DS, Demchinsky AM, Strelnikov VV, Tanas AS, Orlova OM, Machalov AS, Overchenko KV, Markova TV, Golenkova DM, Anoshkin KI, Volodin IV, Zaletaev DV, Pulin AA, Nadelyaeva II, Kalinkin AI, Barh D. Genetic screening of Russian Usher syndrome patients toward selection for gene therapy. Ophthalmic Genet. 2018 Dec;39(6):706-713. doi: 10.1080/13816810.2018.1532527. Epub 2018 Oct 25. PMID 30358468